CLINICAL TRIAL: NCT04131569
Title: Association of Gut Microbiota Diversity With Extended-spectrum Beta-lactamase Producing Enterobacteriales Fecal Carriage and Subsequent Infection in Intensive Care Unit: Microbe Study
Brief Title: Gut Microbiota Association With ESBL-E Colonisation and Subsequent ESBL-E Infection
Acronym: Microbe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bordeaux (Other)
Responsible Party: Principal Investigator, Dr Pauline Esteves, Doctor, University of Bordeaux
Other Study IDs: Microbe
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Extended Spectrum Beta-Lactamase Producing Bacteria Infection; Microbial Colonization; Critical Illness
Keywords: ESBL-E; fecal carriage; microbiota; nosocomial infection
MeSH Terms: conditions — Communicable Diseases; Critical Illness; Cross Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — rectal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESBL-E fecal carriers: Patients with a positive ESBL-E fecal carriage according to routine screening
  Interventions: Diagnostic Test: ESBL-E fecal carriage screening according to routine care
- non ESBL-E fecal carriers: Patients without positive ESBL-E fecal carriage according to routine screening
  Interventions: Diagnostic Test: ESBL-E fecal carriage screening according to routine care

INTERVENTIONS:
Diagnostic Test: ESBL-E fecal carriage screening according to routine care — ESBL-E fecal carriage screening according to routine care

SUMMARY:
Antimicrobial resistance is a major threat worldwide and extended-spectrum beta-lactamase producing Enterobacteriales (ESBL-E) are a leading cause because of their wide dissemination. Gut microbiota seems to be correlated with multi-drug resistant organism carriage. This study thus aims to analyse the correlation between gut microbiota, ESBL-E fecal carriage and subsequent infection.

DETAILED DESCRIPTION:
The rising antimicrobial resistance has led to more than 33,000 deaths in Europe in 2015. Among them, extended-spectrum beta-lactamase-producing Enterobacteriaceae (ESBL-E) are the most frequent in Europe and have disseminated both in the community and in healthcare settings. Some studies have suggested that microbiota could be different between multi-drug resistant organisms, with different relative abundances of some bacteria. One study focused on ESBL-E fecal carriers, but in the community, with Bacteroides uniformis being more abundant in ESBL-E non-carriers than carriers. As identification of species discriminating between ESBL-E fecal carriers and non-carriers could pave the way for the design of ESBL-E carriage eliminating probiotics, we aim to analyse the correlation between gut microbiota and ESBL-E fecal carriage.

Moreover, mechanisms in the link between ESBL-E fecal carriage and subsequent ESBL-E infection remain, so far, poorly understood and this study aims to provide a first insight in the involvement of gut microbiota in the link between colonization and infection.

ELIGIBILITY:
Inclusion Criteria:

* Patient above 18 year-old admitted to intensive care unit
* ESBL-E fecal carriage according to current screening recommendations for ESBL-E carriage group
* Feces quantity on rectal swab adequate for routine screening and microbiota analysis

Exclusion Criteria:

* Guardianship, curatorship, or prisoners
* No health insurance
* No legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every in-patients admitted to our medical intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Gut bacteriobiota diversity according to ESBL specie | at positive screening
  Comparison of gut bacteriobiota alpha diversity between ESBL E. coli and ESBL K. pneumoniae fecal carriers

SECONDARY OUTCOMES:
Gut mycobiota diversity according to ESBL specie | at positive screening
  Comparison of gut mycobiota alpha diversity between ESBL E. coli and ESBL K. pneumoniae fecal carriers
Gut bacteriobiota diversity according to ESBL specie | at positive screening
  Analysis of gut bacteriobiota beta diversity between ESBL E. coli and ESBL K. pneumoniae fecal carriers
Gut mycobiota diversity according to ESBL specie | at positive screening
  Analysis of gut mycobiota beta diversity between ESBL E. coli and ESBL K. pneumoniae fecal carriers
bacteria and the absence of ESBL E. coli fecal carriage | at admission
  Association of bacteria with the absence of ESBL E. coli fecal carriage by LefSe method
fungi and the absence of ESBL E. coli fecal carriage | at admission
  Association of fungi with the absence of ESBL E. coli fecal carriage by LefSe method
fungi and the absence of ESBL K. pneumoniae fecal carriage | at admission
  Association of fungi with the absence of ESBL K. pneumoniae fecal carriage by LefSe method
bacteria and the absence of ESBL K. pneumoniae fecal carriage | at admission
  Association of bacteria with the absence of ESBL K. pneumoniae fecal carriage by LefSe method
Gut bacteriobiota and subsequent ESBL-E infection | at admission
  Comparison of gut bacteriobiota alpha diversity between ESBL-E fecal carriers subsequently ESBL-E infected and non-subsequently ESBL-E infected.
Gut bacteriobiota and subsequent ESBL-E infection | at admission
  Analysis of gut bacteriobiota beta diversity between ESBL-E fecal carriers subsequently ESBL-E infected and non-subsequently ESBL-E infected
Gut mycobiota and subsequent ESBL-E infection | at admission
  Comparison of gut mycobiota alpha diversity between ESBL-E fecal carriers subsequently ESBL-E infected and non-subsequently ESBL-E infected.
Gut mycobiota and subsequent ESBL-E infection | at admission
  Analysis of gut mycobiota beta diversity between ESBL-E fecal carriers subsequently ESBL-E infected and non-subsequently ESBL-E infected
Bacteria and the absence of subsequent ESBL-E infection | at admission
  Association of bacteria with ESBL-E subsequent infection among ESBL-E fecal carriers by LefSe method
Fungi and the absence of subsequent ESBL-E infection | at admission
  Association of fungi with ESBL-E subsequent infection among ESBL-E fecal carriers by LefSe method

OTHER OUTCOMES:
Association of gut bacteriobiota with ventilator-associated pneumonia | at admission
  Patients with oro-tracheal intubation for more than 48 hours among those included will be included in this ancillary analysis. Association of alpha and beta diversities for both gut bacteriobiota and mycobiota with subsequent ventilator-associated pneumoniae will be assessed
Association of gut bacteriobiota with intensive care unit mortality | at admission
  Association of alpha and beta diversities for both gut bacteriobiota and mycobiota with subsequent intensive care unit mortality will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Medical intensive care unit, Pelelgrin hospital, Bordeaux, Nouvelle-Aquitaine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prevel R, Enaud R, Orieux A, Camino A, Sioniac P, M'Zali F, Dubois V, Berger P, Boyer A, Delhaes L, Gruson D. Bridging gut microbiota composition with extended-spectrum beta-lactamase Enterobacteriales faecal carriage in critically ill patients (microbe cohort study). Ann Intensive Care. 2023 Apr 4;13(1):25. doi: 10.1186/s13613-023-01121-0. PMID 37014580